CLINICAL TRIAL: NCT04607759
Title: Randomized Clinical Trial to Analyze the Efficacy of a Supplement Removed From Cucumber on the Articular Pain of Diagnosed Patients of Arthrosis
Brief Title: Clinical Trial on the Articular Pain With a Cucumber Supplement in Patients Diagnosed With Arthrosis
Acronym: CUCART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-00017
Record Dates: First submitted 2020-10-15; First posted 2020-10-29 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (cucumber) (Experimental): Consumption for 90 days of cucumber extract (20mg/day)
  Two capsules a day orally for 90 days.
  Interventions: Dietary Supplement: nutraceutical
- control group Placebo (sucrose) (Placebo Comparator): Two capsules a day orally for 90 days.
  Interventions: Dietary Supplement: nutraceutical

INTERVENTIONS:
Dietary Supplement: nutraceutical — Subjects will consume two capsules for eight weeks

SUMMARY:
Randomized, controlled, double-blind clinical trial of two parallel branches to analyze the efficacy of a supplement extracted from the cucumber on the joint pain of patients diagnosed with osteoarthritis.

DETAILED DESCRIPTION:
The subjects that meet the selection criteria will make a total of two visits to the research laboratory and will carry out the pre-established tests in the protocol. Subsequently, a statistical analysis will be carried out with the variables measured in the study to obtain results.

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years.
* Subjects diagnosed with osteoarthritis with functional grades I-III according to the modified criteria of the American College of Rheumatology.
* Subjects must have persistent knee pain associated with osteoarthritis with a baseline score of at least 30 mm on the VAS pain assessment.
* Subjects should not present narcotic drugs or steroidal anti-inflammatory drugs or immunosuppressants in their treatment.

Exclusion Criteria:

* Serious or terminal illnesses.
* Subjects currently taking glucosamine, chondroitin sulfate, collagen or hyaluronic infiltrations or any supplement indicated for joint health.
* Subjects with chronic inflammatory diseases that affect the musculoskeletal system (rheumatoid arthritis, gout, pseudo-gout, Paget's disease, chronic pain syndrome, etc.).
* Subjects with a body mass index above 32.
* Pregnant or lactating women.
* Inability to understand informed consent.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain from baseline at 8 weeks | The pain will be measured by a scale twice, at the beginning and at the end of the study (after an 8 week consumption).
  Visual analog scale from 0 to 10. The higher the value, the more pain.

SECONDARY OUTCOMES:
Change in concomitant analgesic medication | Twice, once at the beginning of the trial in basal conditions and once at the end after 8 weeks of consumption.
  The change in the need for the use of analgesic medications will be evaluated.
Quality of life test: WOMAC test | it will be measured twice, once at baseline or at the end of the study after 8 weeks of use
  The quality of life of the subjects will be measured with the WOMAC test. It is a 24-item test that will measure the degree of pain: nothing, little, enough, a lot, and a lot, when performing activities in daily life.
Functional test | Twice, once at the beginning of the trial in basal conditions and once at the end after 8 weeks of consumption.
  The balance and mobility of the subjects will be measured with the Timed Up and Go Test
Muscle function | Twice, once at the beginning of the trial in basal conditions and once at the end after 8 weeks of consumption.
  Isokinetic dynamometry.
Inflammatory state IL-b | Twice, once at the beginning of the trial in basal conditions and once at the end after 8 weeks of consumption.
  It is a blood test that measures cartilage degradation
Cartilage metabolism | Twice, once at the beginning of the trial in basal conditions and once at the end after 8 weeks of consumption.
  It is a blood test that measures cartilage degradation
Liver safety variables | Twice, once at the beginning of the trial in basal conditions and once at the end after 8 weeks of consumption.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain